CLINICAL TRIAL: NCT03337945
Title: In Vivo Determination of Cytochrome P450 Activities in Patients With Liver Cirrhosis
Acronym: CombiCapsLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01329
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Liver Cirrhosis
Keywords: CYP450 phenotyping in patients with liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: A single center, single dose, open label, single period study to characterize cytochrome P450 (CYP) isoforms by the use of the Basel Phenotyping cocktail in patients at different stages of liver cirrhosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Basel phenotyping cocktail" capsule (Experimental): Oral intake of "Basel phenotyping cocktail" capsule and pharmacokinetics (PK) sampling
  Interventions: Drug: "Basel phenotyping cocktail" capsule

INTERVENTIONS:
Drug: "Basel phenotyping cocktail" capsule — Oral intake of "Basel phenotyping cocktail" capsule and pharmacokinetics (PK) sampling

SUMMARY:
Subjects will receive the "Basel phenotyping cocktail" capsule orally with 120-200ml tap water in fasted state. After intake peripheral venous blood samples will be drawn.

12 patients (male and female) with liver cirrhosis for each Child Pugh Category A, B, and C, and 12 age- and gender-matched healthy control subjects will be included (in total 48 participants).

ELIGIBILITY:
Inclusion Criteria:

* Full mental and legal capacity.
* Signed informed consent prior to any study related procedure.
* Ability to communicate in German, sufficient to comprehend and adhere to study protocol.
* Normal physical examination, vital signs, laboratory workup, and CombiCaps LC Study Protocol Version 1.2 09.08.2017 Page 9 of 50 electrocardiogram (ECG) (in the opinion of investigator).
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening (in the opinion of investigator).
* No other conditions or circumstances that might interfere with compliance with study protocol (in the opinion of investigator).

Exclusion Criteria:

* Known hypersensitivity to probe substances or any excipient of the drug formulation.
* Ongoing or past treatment with another investigational drug within 30 days prior to screening.
* Concomitant treatment with drugs that inhibit or induce CYP3A4, CYP2D6, CYP2C9, CYP2C19, CYP2B6 and CYP1A2 function (in the opinion of investigator).
* Actual infection
* Severe heart failure (NYHA IV).
* Actual alcohol or drug abuse
* Positive results from urine drug screen at screening.
* Excessive caffeine consumption, defined as >800 mg per day at screening*.
* Subjects unwilling to stop consumption of alcoholic- and caffeine-containing beverages on study days until after the last sampling time-point of the study period.
* Intake of food products (immediately before or during study) known to be inducers or inhibitors of CYP450 (e.g. grapefruit juice)
* Loss of 250 ml or more of blood within 3 months prior to screening.
* Pregnant or lactating women
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening. *100 mg caffeine is approximately 1'000 ml Coca Cola®, 2½ espresso cups or 1 cup of strong coffee.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration-time profile in plasma | -5 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours
  Concentration-time Profiles assessed in Plasma over several time points measuring parent compounds and corresponding metabolites to calculate metabolic ratios

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, Principal Investigator — Universitätsspital Basel, Switzerland
Locations (1):
- Ambulantes Studienzentrum, Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Results of Trial will be published in a peer reviewed Journal

REFERENCES:
- [Derived] Duthaler U, Bachmann F, Ozbey AC, Umehara K, Parrott N, Fowler S, Krahenbuhl S. The Activity of Members of the UDP-Glucuronosyltransferase Subfamilies UGT1A and UGT2B is Impaired in Patients with Liver Cirrhosis. Clin Pharmacokinet. 2023 Aug;62(8):1141-1155. doi: 10.1007/s40262-023-01261-3. Epub 2023 Jun 16. PMID 37328712
- [Derived] Duthaler U, Bachmann F, Suenderhauf C, Grandinetti T, Pfefferkorn F, Haschke M, Hruz P, Bouitbir J, Krahenbuhl S. Liver Cirrhosis Affects the Pharmacokinetics of the Six Substrates of the Basel Phenotyping Cocktail Differently. Clin Pharmacokinet. 2022 Jul;61(7):1039-1055. doi: 10.1007/s40262-022-01119-0. Epub 2022 May 16. PMID 35570253